CLINICAL TRIAL: NCT06253676
Title: Sensing Technologies for Maternal Depression Treatment in Low-Resource Settings
Acronym: StandStrong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Transcultural Psychosocial Organization Nepal (Other); University of Witwatersrand, South Africa (Other); Yale University (Other); Duke University (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Professor of Psychiatry and Behavioral Health, Global Health, and Anthropology, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R33MH126877 (NIH)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Post Partum Depression
Keywords: Low- and Middle-Income Country; Mental Health; Task-Sharing Intervention / Non-Specialist Intervention; mHealth | Digital Health
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Individual-Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor masked to trial arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Delivery of Problem Management Plus (PM+) (Active Comparator): For an eligible, consenting mother participant randomized to the comparator arm, our team will not provide her with active passive sensing technology. As such, no passive sensing data regarding maternal activity and health will be transmitted to or made available to trained, non-specialist providers (i.e., 'PM+ helpers').
  Following enrollment, the mother participant will undergo the five intervention sessions with an assigned PM+ helper in an in-person capacity. In particular, the helper will only deliver the intervention as originally manualized; in other words, s/he will not integrate key findings/interpretations of the aforementioned passive sensing data into delivery.
  Interventions: Behavioral: Problem Management Plus (PM+)
- StandStrong Platform-Informed Delivery of Problem Management Plus (PM+) (Experimental): For an eligible, consenting mother participant randomized to the experimental arm, our team will provide her a smart phone (with EBM application) and her infant with a GPS beacon. Collectively, these passive sensors will non-invasively collect data regarding maternal activity and health (e.g., heart rate, step count, proximity to infant, etc.) from her and the infant. Upon acquisition of said data, we will transmit it to a data analysis engine based in a machine-learning approach and then visualize it within an application (i.e., 'dashboard') available to trained, non-specialist providers (i.e., 'PM+ helpers').
  Following enrollment, the mother participant will undergo the five intervention sessions with an assigned PM+ helper in an in-person capacity. In particular, the helper will integrate key findings/interpretations of the aforementioned passive sensing data into delivery of a given session with respect to an adapted fidelity checklist.
  Interventions: Behavioral: Problem Management Plus (PM+)

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — Validated across multiple low- and middle-income country settings, PM+ is World Health Organization-developed, five-session task-sharing intervention for mild to moderate distress. Per the (manualized) intervention, trained non-specialist providers coach eligible clients to address practical problems and/or distress in their daily lives via the use of fundamental cognitive behavioral strategies (e.g., deep breathing and stress management, behavioral activation, strengthening of social support, etc.).

SUMMARY:
In certain low- and middle- income country settings, there is a disproportionate level of untreated postpartum depression that presents both acute and long-term risks to a mother's well-being. Although there is increasing willingness among health systems to involve non-specialists, such as community health workers, in the delivery of psychosocial interventions for postpartum depression, the effectiveness of these interventions has been mixed. The incorporation of digital technology, though, has the potential to improve the effectiveness of non-specialist-delivered interventions.

The goal of this clinical trial is to evaluate the acceptability and clinical efficacy of the StandStrong intervention- a non-specialist, passive sensing technology-informed (i.e., digital) mental health intervention- as compared to a standard non-specialist mental health intervention among postpartum-depressed mothers in Nepal. Successful completion of the trial will contribute to the optimization of psychosocial intervention delivery for the postpartum context in low- and middle-income country settings.

DETAILED DESCRIPTION:
Among certain low- and middle- income countries, there is a disproportionate level of untreated postpartum depression that presents both acute and long-term risks to a mother's well-being and her child's survival, health, and development. Although there is increasing willingness among health systems to involve non-specialists, such as community health workers, in the delivery of psychosocial interventions for postpartum depression, the outcomes of these interventions have been mixed. Digital technology, specifically the use of passive sensing data collection to quantitatively asses a mother's health and monitor behavior change, has the potential to improve the effectiveness of non-specialist-delivered interventions.

Per this clinical trial, our research team will expand upon previous pilot work and evaluate the StandStrong intervention, a passive sensing technology-informed intervention adapted for postpartum depression. StandStrong- a passive sensing technology platform that consists of passive sensors (i.e., smartphone and GPS beacon), a passive sensing data visualization application, and a passive data analysis engine based in a modern machine-learning approach- transmits passive sensing data from a given mother and her infant to a trained, albeit non-specialist provider who interprets such data and then personalizes the intervention for her. Throughout the trial, the intervention within which this data will be integrated is Problem Management Plus (PM+). Validated across multiple low- and middle-income country settings, PM+ is World Health Organization-developed, five-session task-sharing intervention for mild to moderate distress. Per the (manualized) intervention, trained non-specialist providers coach eligible clients to address practical problems and/or distress in their daily lives via the use of fundamental cognitive behavioral strategies (e.g., deep breathing and stress management, behavioral activation, strengthening of social support, etc.).

In particular, our team will conduct a double-arm, single-blind, individual-randomized controlled trial (RCT) that evaluates the clinical efficacy of platform-informed delivery of the intervention as compared to standard delivery of the intervention. We hypothesize that platform-informed delivery will more significantly reduce severity of symptoms- such as depression, anxiety, and quality of life- associated with postpartum depression relative to standard delivery; moreover, we imagine that platform-informed delivery will prove both cost-effective and scalable. Moreover, we will pose recommendations for platform and intervention implementation within the Nepal health system relative to the RE-AIM framework (i.e., Reach; Effectiveness; Adoption; Implementation; Maintenance).

Successful completion of the trial will contribute to the optimization of psychosocial intervention delivery for the postpartum context in low- and middle-income country settings.

ELIGIBILITY:
Inclusion Criteria:

* Mother Age: 15-39 years
* Infant Age: Within 1st 1000 days of life
* Mother PHQ-9 Score: 8+
* Access to a technology charging modality within home
* Will remain in the study area for a minimum of 6 months after enrollment

Exclusion Criteria:

* Mother PHQ-9 Score: Less Than 8
* Different permanent residences of mother and infant at time of recruitment
* Acute medical need or hospitalization of mother or infant at time of recruitment
* Presentation of psychotic symptoms (as indicated by the psychosis module of the locally validated Community Informant Detection Tool) at time of recruitment

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 20 Weeks Following Baseline Assessment
  9-item self-report scale that assesses severity of depression symptoms
  * Minimum Value = 0
  * Maximum Value = 27
  * Higher scores indicate increased severity of depression symptoms

SECONDARY OUTCOMES:
Psychological Outcome Profiles Questionnaire (PSYCHLOPS) | 20 Weeks Following Baseline Assessment
  4-item self-report questionnaire that indicates a personalized measure of psychological distress
Generalized Anxiety Disorder-7 (GAD-7) | 20 Weeks Following Baseline Assessment
  7-item self-report scale that assesses severity of generalized anxiety symptoms
  * Minimum Value = 0
  * Maximum Value = 21
  * Higher scores indicate increased severity of generalized anxiety symptoms
World Health Organization Disability Assessment Schedule (WHODAS) | 20 Weeks Following Baseline Assessment
  12-item self-report scale that assesses extent of adult disability
  * Minimum Value = 0
  * Maximum Value = 48
  * Higher scores indicate increased severity of disability

OTHER OUTCOMES:
Reducing Tension Checklist | 20 Weeks Following Baseline Assessment
  10-item self-report scale that assesses degree of psychosocial skill use
  * Minimum Value = 0
  * Maximum Value = 30
  * Higher scores indicate increased use of psychosocial skills

CONTACTS AND LOCATIONS:
Overall Officials: Brandon A Kohrt, MD PhD, Principal Investigator — The George Washington University | Center for Global Mental Health Equity
Locations (1):
- Transcultural Psychosocial Organization Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Our research team will make individual participant data available via the National Institute of Mental Health Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Our research team will make data available on or following the trial's award end date.
Access Criteria: Standard access requirements for National Institute of Mental Health Data Archive (NDA)